CLINICAL TRIAL: NCT06647186
Title: Evaluation of Non-Incised Papillae Surgical Approach (NIPSA) Versus Conventional Flap in Periodontal Reconstructive Surgery of Intrabony Defects (Clinical and Radiographic Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bassant Hamdy Mowafey (Other)
Responsible Party: Sponsor-Investigator, Bassant Hamdy Mowafey, Associate professor of Oral Diagnosis and Radiology, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A10020822
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Periodontal Bone Loss
Keywords: Periodontitis; Periodontal regeneration
MeSH Terms: conditions — Alveolar Bone Loss; Periodontitis

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients were randomly selected into either study group (NIPSA) or control group (Conventional falp) using the coin toss method. Hence the study groups were classified into two groups as follows, group I (study group): ten patients treated with NIPSA plus FDBA and group II (Control group): ten patients treated with conventional flap design plus FDBA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Active Comparator): Ten patients treated with Non-Incised Papillae Surgical Approach (NIPSA) plus Allograft bone substitute
  Interventions: Procedure: Non Incised Papillae Surgical Approach
- Control group (Active Comparator): Ten patients treated with Conventional Flap plus Allograft bone substitute
  Interventions: Procedure: Conventional flap design

INTERVENTIONS:
Procedure: Non Incised Papillae Surgical Approach — Ten patients were included in this group, phase I therapy (scaling, root planing and oral hygiene measures) was performed. A single horizontal or oblique incision was made in the mucosa located on the cortical bone tissue, apical to the intrabony defect. The mesiodistal extension of the incision was sufficient to allow access to the defect. Tissue coronal to the incision was raised to full thickness from the incision line to expose the bone peaks delimiting the intrabony defect. The granulation tissue was removed from the bone walls of the defect. Dental plaque and calculus deposits were removed from the root surface with ultrasonic scaler tips and micro-minicurettes. A solution of 24% Ethylenediaminetetraacetic acid (EDTA) was applied to the root surface for 2 min, irrigation with saline solution then allograft bone material was packed into the periodontal defect. The incision was sutured with horizontal internal mattress sutures then simple interrupted sutures.
  Other Names: NIPSA
  Arms: Study group
Procedure: Conventional flap design — Ten patients were included in this group, phase I therapy (scaling, root planing and oral hygiene measures) was performed. Intrasulcular incision was made splitting the buccal papilla from the palatal papilla. All defects were approached by elevating a flap only on the buccal side and leaving the oral portion of the interdental supracrestal soft tissues undetached. The full-thickness elevation of the marginal portion of the flap was performed with a microsurgical periosteal elevator.
  After removal of granulation tissue from the bone walls of the defect, root and defect debridement was performed with manual and mechanical (ultrasonic) instruments with tips for subgingival instrumentation.
  A solution of 24% Ethylenediaminetetraacetic acid (EDTA) was applied to the root surface for 2 min, irrigation with saline solution then allograft bone material was packed into the periodontal defect. The incision was sutured with simple interrupted sutures.
  Other Names: Single flap approach
  Arms: Control group

SUMMARY:
Objectives: To compare the effectiveness of Non-Incised Papillae Surgical Approach (NIPSA) versus conventional flap with mineralized Freeze-Dried Bone Allograft (FDBA) in periodontal reconstructive surgery of intrabony defects (Clinical and Radiographic study).

Patients and methods: Twenty patients with stage III/IV periodontitis with vertical intraosseous defect treated with NIPSA plus FDBA (n=10) or Conventional flap plus FDBA (n=10) were analysed. All patients met the same inclusion criteria and were treated following the same protocol, except for the surgical management of soft tissue (NIPSA versus Conventional flap). Clinical parameters were assessed at baseline, three months and sixmonths. Radiographic parameters were assessed at baseline and six months.

DETAILED DESCRIPTION:
IPatients' selection: Twenty patients with periodontitis were diagnosed with vertical intra-osseous periodontal defects. They were selected from the Department of Oral Medicine and Periodontology, Faculty of Dentistry, Mansoura University putting into consideration certain inclusion and exclusion criteria. The patients have known all of the needed information about the treatment protocols and the materials they would receive. All possible risks and other treatment options had been reviewed and explained to the patients. The patients were cooperative and they understood this explanation. Written consent had been taken from each patient before performing any steps and approved from the ethical committee of our college

Inclusion criteria:

1. Patients with stage III/IV periodontitis.
2. Age Group between 30 to 50 years old.
3. Active residual pockets (positive bleeding on probing) associated with intrabony defects.
4. Periodontal lesions with probing depth (PD) ≥ 5 mm and extension of the intrabony defect ≥ 3 mm.
5. Vertical intrabony periodontal defects, always involving the buccal aspect.

Exclusion criteria:

1. Systemic disease contraindicating periodontal surgery.
2. Smokers.
3. Diabetic patients.
4. Pregnant patients.
5. Third molars or teeth with incorrect endodontic or restorative treatment.

Study Design:

This parallel randomized controlled clinical trial included twenty patients.

The patients selected were classified into two groups:

• Group 1 (Study group): Included ten patients with stage III/IV periodontitis and PD ≥ 5 mm. These patients undergone periodontal treatment using NIPSA procedure in addition to mineralized FDBA substitute for vertical intrabony defects regeneration.

• Group II (Control group): Included ten patients with stage III/IV periodontitis and PD ≥ 5 mm. These patients undergone periodontal treatment using conventional flap procedure in addition to mineralized FDBA substitute for vertical intrabony defects regeneration.

Clinical Periodontal Assessment:

The clinical assessment was performed for all patients at baseline, three and six months after periodontal treatment.

Plaque Index:

It was used to assess the amount of plaque at the gingival third of the tooth. Light source, dental mirrors, sharp dental explorers, periodontal probes and the dryness of the surface of the teeth and gingiva using air were used for scoring the plaque index. Therefore, only the plaque of the cervical third of the tooth was evaluated without regarding extension of the plaque on the middle and incisal thirds.

Gingival Bleeding Index:

The Gingival bleeding index was adopted by Ramfjord to measure the severity of gingivitis and its extension. Measurements of the index were taken from all surfaces of the teeth. A periodontal probe was used for recording the scores from four gingival areas of the tooth which were the distofacial papilla, facial gingival margins, mesiofacial papilla and entire lingual gingival margin of the tooth.

Probing Depth:

Probing depth was measured by special periodontal probe which was (UNC-15 probe). The index focused on how much the periodontal probe went deeper in the periodontal pockets and the reading was taken from the free gingival margin of tooth to the base of the pockets. Measurements were taken from different surfaces per each tooth.

Which were the distofacial surface, mid facial surface, mesiofacial surface, mesio-lingual surface, mid lingual surface and disto-lingual surfaces of the tooth. Adding the six scores per each tooth and dividing it by six gave the mean score for that tooth and to get the index score for the person; the scores for each tooth were added and then were divided by the number of all examined teeth.

Clinical Attachment Loss:

The CAL is the measurement of the distance from a fixed reference point (typically the cemento-enamel junction, CEJ) to the base of the periodontal pocket. It provides valuable information about the extent of attachment loss around teeth. A calibrated periodontal probe (UNC-15) was used to measure probing depth (PD) and calculate CAL. Insert the probe gently into the gingival sulcus or pocket, parallel to the long axis of the tooth, and record the depth from the CEJ to the base of the sulcus or pocket. Measure CAL at multiple sites (e.g., mesial, distal, buccal, lingual) around each tooth to account for variations in attachment loss.

Gingival Recession:

Gingival recession refers to the exposure of the tooth root surface due to the apical migration of the gingival margin. Therefore, gingival recession is associated with the destruction of both soft and hard tissue. It is an important clinical parameter to assess in periodontal evaluations. Gingival recession was measured from the CEJ to the current position of the gingival margin using (UNC-15 probe) inserted gently into the gingival sulcus or pocket, parallel to the long axis of the tooth.

Width of Keratinized Tissue:

Adequate width of keratinized tissue is associated with better periodontal health outcomes, including reduced risk of gingival recession and attachment loss. During periodontal surgeries, adequate keratinized tissue facilitates better wound healing and enhances the success of procedures like gingival grafting. Keratinized tissue width was measured using (UNC-15 probe) from the gingival margin to the mucogingival junction, at the mid-buccal point.

Location of the Tip of the Papilla:

Taking as a reference the central axis of the tooth, the distance from the CEJ in the zenith of the tooth to the vertex of the papilla. The manual UNC-15 probe was used to measure the distance.

Radiographic assessment:

Radiographic interpretation of the intrabony defect was done using CBCT at baseline and 6 months post-operatively. Landmarks were identified using CBCT including the cemento-enamel junction (CEJ), the alveolar crest (AC), the base of the defect (BD) and the depth of intrabony defect (ID).The depth of intrabony defect (ID) was measured as the difference between the distance from (CEJ) to (BD) and (CEJ) to (AC).

V. Surgical Intervention:

Pre surgical phase:

Phase I therapy according to the European Federation of Periodontology (EFP); the S3 Level Clinical Practice Guideline (CPG). The first step in therapy was intended to remove supragingival calculus using ultrasonic scalers and guide behaviour change by encouraging the patient to increase the efficacy of oral hygiene (motivation, oral hygiene instructions) in the form of brushing, flossing, and mouthwash. Prescription of chlorhexidine mouth wash twice daily and the patient was scheduled for a follow-up appointment after 7 days.

The second step of therapy (cause-related therapy) was aimed at controlling (reducing/eliminating) the subgingival biofilm and calculus (subgingival instrumentation) with possible removal of root surface (cementum). Subgingival instrumentation was supplemented with the irrigation of chlorhexidine solution and systemic antibiotic (Metronidazole 500mg) twice daily for 5 days.

All patients were scheduled for a follow-up appointment 2 weeks after step 2 of therapy. The clinical periodontal assessment was re-evaluated to assess if therapy goals were achieved and to verify the eligibility for participating in the study before starting the surgical phase.

Surgical phase:

Group I (NIPSA):

After administration of local anesthesia, using blade number 15, a single horizontal or oblique incision was made in the mucosa located on the cortical bone tissue, apically at the edge of the bone crest that delimited the intrabony defect and as far as possible from the marginal tissues. The mesiodistal extension of the incision was sufficient to allow access to the defect, expose its limits, and allow correct debridement of the periodontal pocket and the application of biomaterials.

Tissue coronal to the incision was raised to full thickness from the incision line to expose the bone peaks delimiting the intrabony defect. In patients with lingual defect, we were able to has a lingual component, the area was accessed using buccal access. The granulation tissue was removed from the bone walls of the defect. Dental plaque and calculus deposits were removed from the root surface with ultrasonic scaler tips and micro-minicurettes.

Group II (Conventional flap):

After administration of local anesthesia, using blade number 15, intrasulcular incision was made splitting the buccal papilla from the palatal papilla. All defects were approached by elevating a flap only on the buccal side and leaving the oral portion of the interdental supracrestal soft tissues undetached. The full-thickness elevation of the marginal portion of the flap was performed with a microsurgical periosteal elevator.

After removal of granulation tissue from the bone walls of the defect, root and defect debridement was performed with manual and mechanical (ultrasonic) instruments with tips for subgingival instrumentation.

Application of bone graft material:

A solution of 24% Ethylenediaminetetraacetic acid (EDTA) was applied to the root surface in all the patients in the two groups, and after 2 min, irrigation with abundant saline solution then allograft bone material; mineralized (FDBA) spongy powder crushed bone preparation of natural cadaver (cadaveric origin) was mixed with sterile saline solution together to produce stable viscous bone graft material then packed into the periodontal defect during surgery.

Suturing technique: NIPSA group: The incision was sutured with a double suture line; the first line with horizontal internal mattress sutures to approximate the connective tissue of the mucosal edges of the incision. The second line with simple interrupted sutures, interrupted sutures help to bring the wound edges together counterbalancing the eversion caused by the horizontal mattress sutures. Conventional group: The incision was sutured with simple interrupted sutures.

Post-operative instructions: All patients received Amoxicillin (Augmentin) 1000 mg every 12h for 5 days. Postoperative pain and inflammation were controlled using ibuprofen (Brufen) 600 mg (or acetaminophen (Doliprane) 1000mg in patients allergic to ibuprofen). Patients rinsed with 0.2% chlorhexidine hydrochloride (Orovex) twice daily for 1 week, without mechanical hygiene on the surgical area.

Statistical analysis of the data Data were fed to the computer and analysed using IBM SPSS software package version 20.0. (Armonk, NY: IBM Corp) Qualitative data were described using number and percent. Shapiro-Wilk test was used to verify the normality of distribution. Quantitative data were described using range (minimum and maximum), mean, standard deviation, median and interquartile range (IQR). Significance of the obtained results was judged at the 5% level.

The used tests were

1. - Chi-square test For categorical variables, to compare different groups.
2. - Student t-test For normally distributed quantitative variables, to compare between two studied groups.
3. - Paired t-test For normally distributed quantitative variables, to compare between two periods.
4. - ANOVA with repeated measures For normally distributed quantitative variables, to compare between more than two periods or stages and Post Hoc Test (adjusted Bonferron) for pairwise comparisons.
5. - Mann Whitney test For abnormally distributed quantitative variables, to compare between two studied groups.
6. - Friedman test For abnormally distributed quantitative variables, to compare between more than two periods or stages and Post Hoc Test (Dunn's) for pairwise comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage III/IV periodontitis.
2. Age Group between 30 to 50 years old.
3. Active residual pockets (positive bleeding on probing) associated with intrabony defects.
4. Periodontal lesions with probing depth (PD) ≥ 5 mm and extension of the intrabony defect ≥ 3 mm.
5. Vertical intrabony periodontal defects, always involving the buccal aspect.

Exclusion Criteria:

1. Systemic disease contraindicating periodontal surgery.
2. Smokers.
3. Diabetic patients.
4. Pregnant patients.
5. Third molars or teeth with incorrect endodontic or restorative treatment.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Gingival Recession | Three and six months

SECONDARY OUTCOMES:
Location of the tip of the papilla | Three and six months
Width of keratenized tissue | Three and six months
Probing depth reduction | Three and six months
Clinical attachment gain | Three and six months
Plaque index | Three and six months
Gingival bleeding index | Three and six months
Bone gain | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Professor Una Mohamed ElShinnawi, Study Chair — Faculty of Dentistry Mansoura University
Locations (1):
- Faculty of Dentistry Mansoura Univesity, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided